CLINICAL TRIAL: NCT01183455
Title: Effect of Intravenous Alpha-1 Antitrypsin on Preserving Beta-cell Function in New-onset Type 1 Diabetes Mellitus (ITN041AI)- Part II
Brief Title: A Research Trial of Aralast NP in New Onset Diabetes (RETAIN) - Part II
Acronym: RETAIN
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision-lack of mechanistic signal and competing industry studies
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAIT ITN041AI Part II
Record Dates: First submitted 2010-08-16; First posted 2010-08-17 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1 (new-onset); T1DM (new-onset); T1D (new-onset); Diabetes, Autoimmune; Alpha1-Proteinase Inhibitor; Alpha-1 Antitrypsin; AAT
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; alpha 1-Antitrypsin Deficiency | interventions — alpha 1-Antitrypsin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aralast NP (Experimental): Participants will receive Aralast NP (90mg/kg) intravenously once a week for 12 weeks.
  Interventions: Drug: Aralast NP
- Placebo (Placebo Comparator): Participants will receive placebo intravenously once a week for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aralast NP — Participants will receive IV infusions of Aralast NP (90mg/kg) once a week for 12 weeks.
  Other Names: Alpha 1-Proteinase Inhibitor Human; Alpha,-antitrypsin; AAT
  Arms: Aralast NP
Drug: Placebo — Participants will receive IV infusions of placebo once a week for 12 weeks.
  Other Names: Placebo for Aralast NP
  Arms: Placebo

SUMMARY:
Aralast NP (alpha-1 antitrypsin, AAT), an alpha-1 proteinase inhibitor (human), was the drug to be tested in this clinical trial. Aralast NP is an anti-inflammatory drug that affects the cells that are thought to be involved in the development of type 1 diabetes mellitus (T1DM, T1D). This study, known as RETAIN, was planned as a two-part trial to investigate the effect of Aralast NP on preserving beta cell function and to determine if the intervention would slow the progression of type 1 diabetes.

Part I of this trial (NCT 01183468) was an open-label, safety and dose level study consisting of two groups. After completion of Part I, including a satisfactory safety review, enrollment in Part II was to begin. Part II was designed as a two-arm, double-blind, placebo-controlled clinical trial, and participants were to be randomly assigned to either the Aralast NP treatment or placebo group.

DETAILED DESCRIPTION:
T1D is an autoimmune disease. This means that your immune system (the part of your body that helps fight infections) mistakenly attacks the cells that produce insulin (beta cells in the pancreas). As beta cells are destroyed by your immune cells, your ability to produce insulin is decreased. Insulin helps keep blood glucose levels normal.

Individuals with T1D who have the ability to produce some of their own insulin (even though they still need to take insulin) may be able to achieve better glucose control than people who produce no insulin at all. Better glucose control has been shown to reduce the long-term complications of diabetes. Previous research has shown that giving medicines to affect the immune system soon after type 1 diabetes is diagnosed may stop, delay or decrease the destruction of beta cells, resulting in better glucose control.

In mouse models of disease, alpha-1 proteinase inhibitors have been shown to reverse new-onset diabetes and induce a state of self-tolerance. The RETAIN clinical trial was intended to investigate the effect of Aralast NP on preserving beta cell function and slowing the progression of T1D.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 1 diabetes (T1D) within the past 100 days
* Positive for at least one diabetes-related autoantibody (anti-GAD; anti-insulin, if obtained within 10 days of the onset of insulin therapy; IA-2 antibody and/or ICA, or ZnT8)
* Peak stimulated C-peptide level greater than (>) 0.2 pmol/mL following a mixed meal tolerance test (MMTT)

Exclusion Criteria:

* Severe active disease (hepatitis, cardiac or pulmonary disease, hypertension, immunodeficiency)
* History of any bleeding or clotting factor deficiencies, or stroke
* History of vascular disease or significant vascular abnormalities
* Positive serology exposure to hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV) or toxoplasmosis
* Clinically active infection with Epstein-Barr virus (EBV), cytomegalovirus (CMV), or tuberculosis (TB)
* Prior or current use of oral, inhaled or intranasal glucocorticoids, or any medication known to cause a significant, ongoing change in the course of T1D or immunologic status
* Prior treatment with alpha1-antitrypsin (AAT) or hypersensitivity to AAT or human plasma-derived products
* Current or prior (within the last 30 days) use of metformin, sulfonylureas, glinides, thiazolidinediones, exenatide, liraglutide, DPP-IV inhibitors or amylin
* Current use of any medication known to influence glucose tolerance (e.g., beta-blockers, angiotensin-converting enzyme inhibitors, interferons, quinidine anti-malarial drugs, lithium, niacin)
* Females who are pregnant or lactating, or are unwilling to defer pregnancy during study participation
* Immunoglobulin A (IgA) deficiency
* Uncontrolled hypertension
* Current life-threatening malignancy
* Any condition that in the investigator's opinion may compromise study participation or may confound the interpretation of the study results

Ages: 8 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Mixed-Meal Tolerance Test (MMTT)-Stimulated 2-hour C-peptide Area Under the Curve (AUC) | Week 52

SECONDARY OUTCOMES:
MMTT-Stimulated Peak and 4-hour C-peptide AUC | Weeks 52 and 104
MMTT-Stimulated 2-hour C-Peptide AUC Assessed Over Time | Weeks 0, 14, 26, 52, and 104
Insulin Use in Units Per Kilogram Body Weight Per Day | Weeks 52 and 104
Hypoglycemic Events Occurring from Randomization to End of Trial | Throughout the Study
Glycosylated Hemoglobin (HbA1c) Levels | Weeks 52 and 104
Emergence of Anti-Alpha 1-Antitrypsin (AAT) Antibodies | Throughout the Study
Frequency and Severity of All Adverse Events (AEs) | Throughout the study
Changes in D-dimer Levels Indicating Alteration in Coagulant/Anticoagulant Balance | Throughout the study
Pharmacokinetic Parameters of Aralast NP | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Weir, MD, Study Chair — Joslin Diabetes Center
Locations (15):
- United States (15):
  - University of California San Diego, La Jolla, California
  - Barbara Davis Center, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - University of Maryland Medical Center, Baltimore, Maryland
  - Calvert Memorial Hospital, Prince Frederick, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - University of Massachusetts Medical School, Worchester, Massachusetts
  - Columbia University, New York, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Hospital of Philadelphia, Philadephia, Pennsylvania
  - Cetero Research San Antonio, San Antonio, Texas

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — http://www.niaid.nih.gov
- See also: Immune Tolerance Network website — http://www.immunetolerance.org
- See also: Juvenile Diabetes Research Foundation (JDRF) — http://jdrf.org/about-jdrf/